CLINICAL TRIAL: NCT01877967
Title: A Randomised Double-blind Placebo-controlled Trial Investigating the Effect of Dietary Supplement VSL#3 on Memory, Attention, Executive Function and Mood in Healthy Older Adults.
Brief Title: Investigating the Effect of Dietary Supplement VSL#3 on Cognition and Mood in Healthy Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Actial Farmaceutica S.r.l. (Industry)
Responsible Party: Principal Investigator, Prof. Brian Lawlor, Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 8AA.N04022
Record Dates: First submitted 2013-05-22; First posted 2013-06-14 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Alteration of Cognitive Function; Disturbance in Affect (Finding)
MeSH Terms: conditions — Signs and Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): This group will intake the recommended daily amount of the food supplement VSL#3 (two sachets of the supplement in powder form) every day for twelve weeks. The two sachets will either be taken together or one in the morning and one in the evening.
  Interventions: Dietary Supplement: VSL#3
- Placebo (Placebo Comparator): This group will intake two sachets (2x4.4g) of a placebo each day for 12 weeks. The placebo is in the same powdered form as the food supplement taken by the intervention group. The two sachets will either be taken together or one in the morning and one in the evening.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 — The intervention group will be asked to ingest two sachets (2x4.4g) of the food supplement (VSL#3) each day for 12 weeks, either both at the same time, or one in the morning and one in the evening. This food supplement is in powder form and can be ingested with either cold food or any non-carbonated cold drink. The control group will be given a placebo, although as it is a double-blind intervention, will not know it is a placebo. They will similarly to the intervention group be asked to take two sachets (2x4.4g) of a powder rach day for 12 weeks, either both at the same time, or one in the morning and one in the evening.
  Arms: Intervention
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
This research aims to determine whether a 12 week daily dose of VSL#3 has any measurable effects on memory, attention, executive function or self-reported mood and anxiety in healthy older adults.

DETAILED DESCRIPTION:
This research aims to investigate the effect of dietary supplement VSL#3 on memory, attention, executive function and mood in healthy older adults.

The study will be a randomised double-blind placebo-controlled design and eighty participants will be recruited to take part. Forty participants will be randomly allocated to the food supplement and 40 to placebo. As the sample is initially self-selecting where individuals volunteer to take part, a minimisation procedure will be used to randomise group allocation (Altman & Bland, 2005), with volunteers stratified by gender. Neither the participant nor the research assistant supplying the supplement will know which preparation is administered, thus ensuring double-blind administration.

Participants will be asked to take the food supplement daily for 12 weeks and the pre- and post- intervention data will be collected immediately before and after this time period.

Both pre- and post-intervention data will be collected using validated neuropsychological measures, cognitive measures, EEG and self-report questionnaires. Blood sampling will be conducted pre- and post-intervention by a Research Assistant trained in phlebotomy. Analysis will be carried out on each of the measures using a two-way ANCOVA, using the pre-treatment score as covariate.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 65 and 75
* MMSE score > 23
* Willingness to give informed consent
* Commitment to take the VSL#3 supplement daily for 12 weeks
* Alcohol consumption less than 21 units per week (men), 14 units per week (women)

Exclusion Criteria:

* Current psychoactive medication
* Significant active medical conditions
* History of major psychiatric or neurological condition
* Smoker
* History of epilepsy
* History of traumatic brain injury
* History of immunodeficiency
* Taking immunosuppressants or corticosteroids

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Changes in cognition | Pre and Post the 12 week Intervention
  Measures used to assess cognition:
  Mini Mental State Exam National Adult Reading Test Free and Cued Selective Reminding Test (FCSRT) Category Fluency Task (Animal Fluency) Colour Trials test 1 & 2 Sustained Attention Response Task Choice Reaction Time Task Prospective Memory Task Self-Rated Memory Electrophysiological Measures (EEG spectral power - alpha range 8-14Hz)

SECONDARY OUTCOMES:
Changes in Mood | Pre and Post the 12 week Intervention
  Measures used to assess changes in mood:
  Centre for Epidemiologic Studies Depression Scale (CES-D) Hospital Anxiety and Depression Scale - Anxiety Scale (HADS-A)

OTHER OUTCOMES:
Changes in levels of elements in blood | Pre and Post the 12 week Intervention
  Blood samples will be taken by a Research Assistant trained in Phlebotomy and tested for the presence of homocysteine, folate and vitamin B12 levels, PCR, glucose, insulin, ceramide and metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lawlor, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Institute of Neuroscience, Trinity College, Dublin, Dublin, Co. Dublin, Ireland

REFERENCES:
- [Background] Altman DG, Bland JM. Treatment allocation by minimisation. BMJ. 2005 Apr 9;330(7495):843. doi: 10.1136/bmj.330.7495.843. No abstract available. PMID 15817555